CLINICAL TRIAL: NCT06131814
Title: Comparative Effects of Integrated and Isolated Resisted Exercise on Strength, Power and Endurance in Gym Beginners
Brief Title: Effects of Integrated And Isolated Resisted Exercise on Strength, Power And Endurance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/2023
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Integrated Resisted Training; Isolated Resised Training
Keywords: Endurance; Gym Beginner; isolated training; integrated resisted training; power; resisted exercise; strength training

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail
Who Masked: Outcomes Assessor
Masking Description: Assessor who will take the resdings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): :- The INT program will involve a standard warm-up and cool down. The INT program involve exercises aimed at improving core stability, power, and strength. These exercises will progressed to more demanding exercises over the 8-week training program. The intensity increased by adding more repetitions, resistance, and through exercise modifications. Integrated resisted exercises include opposite arm and leg lift, bridging, side lying lift, ball back extension, push up 5 times repetition twice a week in first 4 week and then progress to 10 times repetition twice a week from 5-8th week of session
  Interventions: Other: 2 groups
- Group 2 (Experimental): The ISO program involved participants first performing a series of standardized warm up and cool down exercises before and after the training program, respectively. Specifically, the participants rode a stationary bike for 10 minutes followed by static stretching of the calves, hip flexor, and low back. The ISO program began with 5 time repetition and lower body resistance exercises for the first 4 weeks and progressed to 10 exercises for the last 4 weeks. The exercise resistance used in the ISO program also progressed over the 8 weeks. The static stretches were repeated as part of the cool down after completing the ISO program. Isolated exercises include leg press, bench press, Ab crunch, barbell curl and back squat
  Interventions: Other: 2 groups

INTERVENTIONS:
Other: 2 groups — up 5 times repetition twice a week in first 4 week and then progress to 10 times repetition twice a week from 5-8th week of session
  Other Names: integrated Resised Training; Isolated resisted training

SUMMARY:
Resistance training and strength training are synonymous terms used to denote a component of sport and exercise training that is designed to enhance muscular strength, muscular power, and local muscular endurance for general exercise or competitive sports. Resistance training is a specialized method of conditioning that involves the use of different modes of training with a wide range of resistive loads, from body weight to barbells. Resistance-training programs may include the use of free weights (barbells and dumbbells), weight machines, medicine balls, kettlebells, elastic tubing, or a person's own body weight to provide the resistance needed to increase strength.

Objective of study is to compare the effects of integrated and isolated resisted exercise on strength, power and endurance in gym beginners. Design of the study is randomized clinical trial. Data will be collected from body choice gym township, Lahore. Performance, strength, power and endurance will be measured by using Borg Rating of Perceived Exertion (RPE) scale, 1RM maximum, Anthropometry. One Group participants will received integrated resisted training session and other group will train with isolated resisted training.

DETAILED DESCRIPTION:
The objective of this study is to compare the effects of integrated and isolated resisted exercise on strength, power and endurance in gym beginners.Resistance training is one of the most popular training approaches adopted by coaches professionals. Due to the limited number of literature on athletes, it's forever a challenge for physiotherapists in to enhance functional performance in players by implementing these techniques.

The basic purpose of this research is to find and compare the effects of integrated and isolated training on strength, power and endurance in gym beginner. The study can help coaches and trainers to identify the most effective training methods for improving strength, power and endurance.Previous literature show that resisted exercises play effective role in gym trainer for strengthening, power and endurance. But there is a limited literature on comparing the effects of integrated and isolated resisted exercise so our focus is to measure the role of these techniques for strength, power and endurance in gym beginners.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18-30 years

  * Male gender only
  * Participants join the gym having duration less than 6 months

Exclusion Criteria:

* Engaged in regular exercise program within the past 6 months

  * History of lower limb injuries or surgeries within the past 6 months
  * Chronic diseases that affect physical function, such as cardiovascular disease, diabetes, or neurological disorders

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male gender only
  • Participants join the gym having duration less than 6 months
Enrollment: 54 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Endurance: sit up test | 1-8 weeks
  The sit-up test is a measure the endurance of the abdominal and hip-flexor muscles. The aim of this test is to perform as many sit-ups as you can in two minutes
Power: - vertical Jump Test | 1-8 weeks
  The person puts chalk on their finger tips to mark the wall at the height of their jump. The person then stands away from the wall, and jumps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump
Strength: 1RM maximum | 1-8 weeks
  The 1RM test is often considered the 'gold standard' for assessing the strength capacity of individuals. It is simply defined as the maximal weight an individual can lift for only one repetition with correct technique

CONTACTS AND LOCATIONS:
Overall Officials: Dr Usama Tahir Butt, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- PSB-Coaching Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hilkens L, Cruyff M, Woertman L, Benjamins J, Evers C. Social Media, Body Image and Resistance Training: Creating the Perfect 'Me' with Dietary Supplements, Anabolic Steroids and SARM's. Sports Med Open. 2021 Nov 10;7(1):81. doi: 10.1186/s40798-021-00371-1. PMID 34757466
- [Background] Saeterbakken AH, Chaudhari A, van den Tillaar R, Andersen V. The effects of performing integrated compared to isolated core exercises. PLoS One. 2019 Feb 27;14(2):e0212216. doi: 10.1371/journal.pone.0212216. eCollection 2019. PMID 30811444
- [Background] Herold F, Torpel A, Schega L, Muller NG. Functional and/or structural brain changes in response to resistance exercises and resistance training lead to cognitive improvements - a systematic review. Eur Rev Aging Phys Act. 2019 Jul 10;16:10. doi: 10.1186/s11556-019-0217-2. eCollection 2019. PMID 31333805
- [Background] Radwan NL, Mahmoud WS, Mohamed RA, Ibrahim MM. Effect of adding plyometric training to physical education sessions on specific biomechanical parameters in primary school girls. J Musculoskelet Neuronal Interact. 2021 Jun 1;21(2):237-246. PMID 34059568
- [Background] Lee SY, Goh A, Tan K, Choo PL, Ong PH, Wong WP, Wee SL. Effectiveness of a community-delivered pneumatic machine resistance training programme (Gym Tonic) for older adults at neighbourhood senior centres - a randomized controlled trial. Eur Rev Aging Phys Act. 2021 Oct 7;18(1):21. doi: 10.1186/s11556-021-00273-x. PMID 34620081
- [Background] Marcos-Pardo PJ, Orquin-Castrillon FJ, Gea-Garcia GM, Menayo-Antunez R, Gonzalez-Galvez N, Vale RGS, Martinez-Rodriguez A. Effects of a moderate-to-high intensity resistance circuit training on fat mass, functional capacity, muscular strength, and quality of life in elderly: A randomized controlled trial. Sci Rep. 2019 May 24;9(1):7830. doi: 10.1038/s41598-019-44329-6. PMID 31127163